CLINICAL TRIAL: NCT02441660
Title: Capsaicin 8% Patch for Spinal Cord Injury Neuropathic Pain
Acronym: Capsaicin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HSC20150322H
Record Dates: First submitted 2015-04-28; First posted 2015-05-12 (Estimated); Results first posted 2022-10-06 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Spinal Cord Injuries; Neuropathic Pain
MeSH Terms: conditions — Spinal Cord Injuries; Neuralgia | interventions — Capsaicin; Transdermal Patch

STUDY DESIGN:
Intervention Model Description: Study participants are assigned to both strengths of the intervention, so all study participants receive both strengths, thus acting as their own control. Data will be compared according to intervention, rather than following each subject from beginning of study through both interventions.
Who Masked: Participant

ARMS (2):
- Investigational Capsacin, Then Control Capsacin (Experimental): Qutenza, Capsaicin 8% Patch will be used for 12 weeks followed by capsacin 0.025% Well Patch
  Interventions: Drug: Capsaicin 8% Patch; Drug: Low Dose Capsaicin 0.025% Well Patch
- Control Capsacin, Then Investigational Capsacin (Experimental): Active control with low dose capsaicin 0.025% Well Patch used for 12 weeks followed by Qutenza 8% Patch
  Interventions: Drug: Capsaicin 8% Patch; Drug: Low Dose Capsaicin 0.025% Well Patch

INTERVENTIONS:
Drug: Capsaicin 8% Patch — Applied topically for 1 hour
  Other Names: Qutenza
Drug: Low Dose Capsaicin 0.025% Well Patch
  Other Names: Control Capsacin patch

SUMMARY:
A prospective case control study to determine the effectiveness and longevity of 8% capsaicin patch(es) in treating neuropathic pain in persons with spinal cord injury. The investigators will study spinal cord injury patients at South Texas Veterans Health Care Systems Spinal Cord Injury inpatient unit and outpatient clinics.

DETAILED DESCRIPTION:
The investigators will recruit ~ 20 patients with chronic spinal cord injury (SCI) and chronic neuropathic pain (>6months) below level of injury who have failed multiple pharmacological agents. Pre-study data collection will include subjective description of pain, baseline visual analog scale (VAS), numeric pain rating scale (NPRS), a numerical scale such as short form (SF) 36 form that measures quality of life parameters, subjective functional independence (FIM) scores, and pain diagrams will be obtained on each participant. Written informed consent will be obtained. After randomization patients will be assigned to a different sequence of treatment.

All patients will receive either the treatment and control patches in a randomized order for a total of three treatment periods (control, treatment, treatment for example). When assigned to received treatment arm of study patients will receive Qutenza Capsaicin 8% patch(es) applied for 1 hour after pre- treatment with topical lidocaine. The control group will receive a low dose (0.04%) amount of capsaicin in patch form using an identical application procedure.

Investigators will give each patient a diary to self record daily VAS/NPRS scores. Investigators will then schedule routine f/u via telephone call at 2, 4, 8, and 12 weeks post application to accurately report onset of relief and obtain NPRS scores at 2, 4, 8, 12 week points. Patients will follow up in clinic at the end of the 12 week study to repeat data collection using our quality of life scale (SF 36) and FIM scores. Investigators will then use data analysis to record percentage of reduction in NPRS/ VAS, and changes in SF 36 and FIM scores at any given time point vs baseline. For those that continue to have pain relief at 12 week mark we will periodically call every 4 months after study completion to assess for total duration of pain relief for up to 1 year post application.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of SCI
2. Neuropathic pain below level of injury
3. Surface area of pain no larger than 2 patches
4. Failed or did not tolerate gabapentin 3600mg/day, pregabalin 600mg/day, capsaicin cream and/or lidocaine cream
5. Skin over painful area intact

Exclusion Criteria:

1. Pain over open wound
2. Previously documented allergy to capsaicin
3. Superficial burn over area of pain
4. Premorbid (before SCI) neuropathic pain
5. HIV/AIDS neuropathy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-04; Primary Completion 2021-07-31 (Actual); Study Completion 2022-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Trbovich, MD, Principal Investigator — South Texas Veterans Health Care System
Locations (1):
- Audie Lee Murphy VA Hospital, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants will be randomized to either the low dose control capsacin or the higher dose 8% capsacin intervention first, and after 12 weeks, will be assigned to the opposite intervention for 12 weeks so that each person acts as their own control. Data collected will compare only the investigational drug group to the control group.
Groups:
- Qutenza Patch Followed by Low Dose Control Patch: The 8% Qutenza patch will administered for 12 weeks followed by the low dose control patch for 12 weeks
- Control Patch, Then Qutenza Patch: The Low dose control patch will administered for 12 weeks followed by the 8% Qutenza patch for 12 weeks
Period: Sequence 1 (12 Weeks)
Arm/Group | Qutenza Patch Followed by Low Dose Control Patch | Control Patch, Then Qutenza Patch
Started | 5 | 6
Completed | 5 | 6
Not Completed | 0 | 0
Period: Sequence 2 (12 Weeks)
Arm/Group | Qutenza Patch Followed by Low Dose Control Patch | Control Patch, Then Qutenza Patch
Started | 5 | 6
Completed | 5 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study Demographics: All subjects were included in both arms of the study, so demographics are reported together for all participants.
Arm/Group | Overall Study Demographics
Number analyzed (Participants) | 11
Age, Continuous [Mean (Full Range); unit: years] | 49.72 [32 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Relief With Visual Analog (VAS) Pain Scale
Description: The Visual Analog Scale (VAS) was used as the primary outcome measure to quantify pain on a scale of 0-10, with 0 being no pain and 10 being the worst pain. VAS was measured at weeks 2,4,6,8,10 and12 during each 12- week block.
Time Frame: Change in pain at 2,4,6,8, 10 and 12 weeks
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Experimental Group: Qutenza, Capsaicin 8% Patch will be used
  Capsaicin 8% Patch: Applied topically for 1 hour
- Control Group: Active control with low dose capsaicin
  Low Dose Capsaicin 0.04% gel
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 11 | 11
score on a scale
  2 weeks | 3.586 (0.5345) | 5.494 (0.5775)
  4 weeks | 4.041 (0.5345) | 5.677 (0.5345)
  6 weeks | 4.984 (0.5540) | 5.768 (0.5345)
  8 weeks | 4.184 (0.5540) | 4.834 (0.5544)
  10 weeks | 4.284 (0.5540) | 4.753 (0.5769)
  12 weeks | 4.049 (0.5775) | 4.311 (0.6795)

2. Primary Outcome: Change in Quality of Life as Measured by the World Health Organization Quality of Life (WHOQOL-BREF)
Description: The World Health Organization Quality of Life (WHOQOL-BREF) questionnaire is a scale used to assess an individual's perception of their quality of life. Its domains include physical health, psychological health, social relationships, and patient environment. It is scored from 0-100, where lower scores indicate poorer perception of quality of life and higher scores indicate better perception. This scale was used to investigate if there was any pattern of change in QOL due to improved pain control. WHO-QOL-BREF was also measured every 4 weeks of each period.
Time Frame: Every 4 weeks for 12 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 11 | 11
score on a scale
  4 weeks | 79.26 (4.092) | 80.91 (4.092)
  8 weeks | 80.91 (4.204) | 85.42 (4.207)
  12 weeks | 74.90 (4.092) | 87.42 (4.207)

3. Primary Outcome: Change in Spinal Cord Independence Measure (SCIM)
Description: The Spinal Cord Independence Measure (SCIM) is a reliable scale that measures proficiency of activities of daily living (ADL's) of patients with spinal cord injuries. (28) It is broken up into four subscales including self-care, respiration and sphincter control, and mobility with a total score combining all 3 outcomes.
  It is scored from 0-100, where lower numbers indicate more dependence on others and higher numbers indicate less dependence. This tool can be applied practically to the study to investigate everyday function before and after patch application. SCIM was administered every 4 weeks of each period.
Time Frame: Every 4 weeks for12 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 11 | 11
score on a scale
  4 weeks | 20.32 (0.9886) | 18.86 (0.9886)
  8 weeks | 20.70 (1.0132) | 18.66 (1.0140)
  12 weeks | 19.23 (0.9886) | 18.86 (1.0140)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Baseline to 24 weeks at the end of treatment to include both experimental and control group assignment.
Arm/Group | Experimental Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-24): https://cdn.clinicaltrials.gov/large-docs/60/NCT02441660/Prot_SAP_000.pdf